CLINICAL TRIAL: NCT05603468
Title: Effect of Platelet-Rich Plasma vs Corticosteroid Injection in Distinct Rotator Cuff Tendinopathy Subtypes in Arthroscopic Repair: a Multicenter, Three-group, Randomized Controlled Trial
Brief Title: Effect of PRP vs Corticosteroid in Rotator Cuff Tendinopathy Subtypes in Arthroscopic Repair
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0833
Record Dates: First submitted 2022-10-25; First posted 2022-11-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Tendinopathy
Keywords: Tendinopathy; Platelet Rich Plasma
MeSH Terms: conditions — Tendinopathy | interventions — Adrenal Cortex Hormones; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet Rich Plasma group (Experimental): patients rejected with platelet rich plasma
  Interventions: Drug: platelet rich plasma
- Corticosteroid group (Active Comparator): patients rejected with corticosteroid
  Interventions: Drug: Corticosteroid
- Normal saline group (Placebo Comparator): patients rejected with normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: platelet rich plasma — Platelet rich plasma group: after the surgery of rotator arthroscopic rotator cuff repair, 3ml PRP (LongTai Biological Company) was injected into the rotator cuff tear under the rotator arthroscope for a time. PRP production process: before anesthesia, 20ml arterial blood was drawn and injected into the PRP tube. The blood was fully oscillated in the tube, and then placed in a centrifuge with 1500g for 9min to remove excess plasma and make 5ml PRP. 3ml is used for injection and 2ml is used for quality control.
  Arms: Platelet Rich Plasma group
Drug: Corticosteroid — Corticosteroid group: after the surgery of rotator cuff repair under arthroscopy, 1mL prednisone (MSD) + 2mL sodium hyaluronate (biochemical Industry Co., Ltd.) was injected under arthroscopy.
  Arms: Corticosteroid group
Drug: Normal saline — Normal saline
  Arms: Normal saline group

SUMMARY:
Prospective, multicenter, randomized, single-blinded, parallel group，placebo-controlled，three-group establishment of specific treatment regimen for subtypes of tendinopathy

DETAILED DESCRIPTION:
This clinical trial uses machine learning to match molecular and clinical features，so as to establish a "rapid recognition system of tendinopathy subtypes" and compares the clinical effects of corticosteroid，platelet rich plasma or placebo on different subtypes of tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff tears were diagnosis by magnetic resonance imaging or arthroscopy
* Surgical intervention of rotator cuff tears was proposed.
* Simple full-layer tear of supraspinatus tendon.
* Patients give informed consent, and sign the informed consent form, and the process must meet the requirements of GCP

Exclusion Criteria:

* Patients with rotator cuff injuries involving infraspinatus, subscapularis, and teres minor tendon injuries
* Patients platelet concentration is lower than 100×109
* Patients have other shoulder diseases, including osteoarthritis, cervical spondylosis, etc.patients have inflammatory diseases, including rheumatoid arthritis, fibromyalgia, rheumatic polymyalgia, etc.patients have received injection treatment within 3 months.
* Patients have participated in clinical trials or are conducting other clinical trials within 3 months before screening.
* Patients have severe primary cardiovascular disease, lung disease, endocrine and metabolic disease or serious diseases that affect their survival, such as tumor or AIDS, the researchers believe that it is not suitable to be selected.
* Patients have severe liver, kidney and hematological lesions, such as kidney function exceeding the upper limit of normal value and liver function exceeding 2 times the upper limit of normal value.
* Patients have viral hepatitis, infectious diseases, severe abnormalities in blood coagulation and other diseases that the researchers consider unsuitable for surgery.
* Women who are pregnant or lactating, or who plan to conceive during follow-up, those who are positive for human chorionic gonadotropin before sampling; menstrual women should wait for surgery after the end of menstruation.
* Patients have severe neurological and mental disorders.
* Patients suspect or do have a history of alcohol or drug abuse.
* Patients have height body mass index (BMI) > 30.
* Patients have tendon disease caused by systemic immune or other diseases, and patients with diseases or symptoms that may affect pain or function scores.
* Patients have coagulation disorders caused by any other acute or chronic disease.
* MRI detection of contraindications. Include, but are not limited to: installation of pacemakers, defibrillators, cardiac stents, artificial heart valves, metal clips after aneurysm surgery, drug infusion devices implanted in the body, any electronic devices implanted in the body (nerve stimulators, bone growth stimulators), endovascular embolization steel rings, filters, ECG recording monitors, metal sutures, shrapnel or iron particles in the body, fixation of steel plates and nails after fracture surgery, Cochlear implant, middle ear graft, intraocular metal foreign body, etc. Claustrophobia, critically ill patients, etc.
* Refer to the April 2008 edition of the Law of the people's Republic of China on the Protection of disabled Persons, patients belong to the subjects of legal disabled persons
* Other situations in which the researchers judged that the subjects were not suitable to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score (OSS) | 6months after surgery
  The Oxford Shoulder Score (OSS) consists of 12 questions with five options each. The light to heavy lines were assigned 1, 2, 3, 4 and 5 points respectively. So the total score is between 12 and 60. A score of 12 represents perfectly normal shoulder function and a score of 60 represents the most severe difficulty in shoulder function.

SECONDARY OUTCOMES:
Oxford Shoulder Score (OSS) | 3 months, 1year, and 2years after surgery
  The Oxford Shoulder Score (OSS) consists of 12 questions with five options each. The light to heavy lines were assigned 1, 2, 3, 4 and 5 points respectively. So the total score is between 12 and 60. A score of 12 represents perfectly
Constant-Mulery score(CMS) | 3 months, 6months, 1year, and 2years after surgery
  The Constant-Mulery score mainly includes 8 aspects related to your shoulder in the past 4 weeks.
  The proportion of subjective and objective components in the Constant-Mulery score is 35 points/65 points. A total of 100 points.The subjective part of the score includes the score of pain degree and the score of impact on daily life. 35 points in total.The objective part of the score includes the score of shoulder range of motion and strength. 65 points in total.
Fear-avoidance belief questionnaire(FABQ) | 3 months, 6months, 1year, and 2years after surgery
  The FABQ is a self-assessment scale with 16 options. Each option has 0~6 points and 7 grades (from extremely disagreeable to extremely agreed). "0" means completely disagreed, "6" means completely agreed, and "1~5" means not sure. The higher the score, the more inclined to fully agree.
Insomnia Severity Index(ISI) | 3 months, 6months, 1year, and 2years after surgery
  The scale is a simple tool for screening insomnia, including 7 items, which are used to evaluate the nature and symptoms of sleep disorders of subjects.
Hospital Anxiety and Depression Scale(HADS) | 3 months, 6months, 1year, and 2years after surgery
  HADS is a self-assessment scale, including two subscales, HADS-A and HADS-D, with a total of 14 items, including 7 items for anxiety (A) and 7 items for depression (D). Each item is scored at four levels according to the frequency of symptoms in the past month. Each item is scored at 0-3 points in four levels. The higher the score, the more serious the anxiety or depression.
SF-36 | 3 months, 6months, 1year, and 2years after surgery
  SF-36 is a concise health questionnaire developed by the Boston Institute of Health, which is widely used in the measurement of the quality of life of the general population, the evaluation of clinical trials and the evaluation of health policies. SF-36 is used to assess physiological function, physiological function, physical pain, general health, energy, social function, emotional function and mental health, which are classified into "physical health" and "mental health"
Visual analogue scale(VAS) | 3 months, 6months, 1year, and 2years after surgery
  Draw a 10cm horizontal line on the paper. One end of the line is "0", indicating no pain; the other end is "10", indicating severe pain; The middle represents different degrees of pain; Let the patient draw a mark on the horizontal line according to their feelings to indicate the degree of pain.
range of motion | 3 months, 6months, 1year, and 2years after surgery
  Measure the patient's flexion, abduction, internal rotation and external rotation angle
muscle strength | 3 months, 6months, 1year, and 2years after surgery
  Use dynamometer to evaluate patient's forward bending, abduction, external rotation and internal rotation strength.
retear rate | 3 months, 6months, 1year, and 2years after surgery
  Proportion of the total number of people with retearing after arthroscopic rotator cuff repair
Acromiohumeral distance | 3 months, 6months, 1year, and 2years after surgery
  Measurement of acromiohumeral distance based on x-ray
Signal to noise ratio of tendon in MRI | 3 months, 6months, 1year, and 2years after surgery
  Measurement of Signal to Noise Ratio of Tendon in MRI based on software

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China